CLINICAL TRIAL: NCT04323020
Title: CT Perfusion (CTP) for Assessment of Poor Neurological Outcome in Comatose Cardiac Arrest Patients (CANCCAP)-a Prospective Cohort Study
Brief Title: CT Perfusion (CTP) for Assessment of Poor Neurological Outcome in Comatose Cardiac Arrest Patients
Acronym: CANCCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Medical Service Foundation (Other)
Responsible Party: Principal Investigator, Jai Shankar, Professor, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS23646 (B2020:017)
Record Dates: First submitted 2020-03-17; First posted 2020-03-26 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Cardiac Arrest
Keywords: Comatose cardiac arrest patients; Computed Tomographic Perfusion; Targeted Temperature Management; Out of hospital cardiac arrest
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Masking Description: Participant will be comatose cardiac arrest
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comatose cardiac arrest patients (Experimental): Comatose cardiac arrest patients will be undergoing CT perfusion test
  Interventions: Diagnostic Test: CT Perfusion

INTERVENTIONS:
Diagnostic Test: CT Perfusion — CT Perfusion

SUMMARY:
ABSTRACT

Brief Overview: Neurological assessment of comatose cardiac arrest patients (CCAP) is challenging because most of these patients are treated with sedatives and therapeutic hypothermia that prevent complete neurological/clinical assessment. A complete and reliable neurological assessment is needed for patient's long-term function and survival. A poor-quality clinical assessment results in resource-intensive treatment that may not benefit the patient. An ancillary test of head CT scan is often used for additional information. However, this additional information still limits the quality of the assessment. In a small pilot study, we explored an advanced CT scan of brain called CT Perfusion (CTP) relative to clinical assessment in CCAP as a predictor of neurological outcome (severe disability or death) at hospital discharge. The preliminary results suggested that CTP was both valid and reliable, relative to clinical assessment, while meeting many of the criteria of an ideal test (fast, safe, accessible, valid, reliable). This project aims to carry out a fully powered study to confirm these findings.

The goal of this project is to validate CTP for predicting neurological outcome at hospital discharge in CCAP. We will conduct a prospective cohort study to validate the use of CTP in CCAP.

Hypothesis- Computed Tomographic Perfusion (CTP) can reliably diagnose potentially fatal brain injury in CCAP in early stage upon hospital admission, which may or may not be recognized in the usual clinical practice due to inadequate clinical examination.

Primary Objective: To validate CTP, relative to the reference standard of clinical assessment, for characterizing poor neurological outcome at hospital discharge in CCAP.

Secondary Objectives:

To establish the safety and inter-rater reliability of CTP in CCAP.

DETAILED DESCRIPTION:
This study will be conducted in our tertiary care cardiac center. The cohort will consist of newly admitted comatose adults (>18 years of age) who have suffered an OHCA and are treated with standard TTM to 36°C. Just before admission to the intensive care unit (ICU), CCAP undergo CT scan of head. Our plan is to add CTP of whole head at the time of their standard of care CT scan of head. CCAP will then be transferred to ICU for further standard management including TTM.

Immediately after acute care, CCAP usually undergo a CT scan of the head, as per standard protocol, to assess for any intracranial pathology. CTP will be performed at the same time as this standard-of-care CT scan of head. CTP images will be acquired according to a standardized stroke imaging protocol in order to ensure whole brain coverage. The CTP data will be transferred to the study imaging core lab at the department of Radiology, University of Manitoba, Winnipeg for interpretation. The CTP results will not be available to the treating physicians and the routine care of the patient will continue as per local practice.

CTP analysis will be performed in the imaging core lab using a semiautomatic deconvolution algorithm on a vendor neutral software package. CTP will be assessed both quantitatively as well as qualitatively.

* Quantitative assessment: Brain death will be defined as CBF <5 mL/100g/min and CBV <2 mL/100g in the brainstem.
* Qualitative assessment: Brain death will be defined as matched decrease of CBF and CBV in the brainstem. The perfusion maps for CBF and CBV will be assessed for binary outcome of 'dead' or 'not-dead', according to our previously published methods.

The perfusion maps will be assessed by the two independent neuroradiologists, who are blinded to each other's assessment and to the clinical history of each patient. If the two neuroradiologists disagree, a consensus agreement will be achieved for the final analysis. Consensus decision reflects the real-life scenario faced in such situations. CTP parameters (CBF and CBV) will be qualitatively assessed for the presence or absence of matched decrease of CBF and CBV.

ELIGIBILITY:
Inclusion Criteria:

* Newly admitted comatose adults (≥18 years old) who have suffered an Out of Hospital Cardiac Arrest (OHCA)
* Treating physicians plan on instituting post cardiac arrest Targeted Temperature Management (TTM) therapies

Exclusion Criteria:

* No substitute decision maker available for consent
* Known pregnancy
* Known contraindication to CT contrast agent, such as a history of allergy or anaphylactic reaction
* Known chronic kidney disease, stage 4-5 (eGFR < 30 mL/min/1.73 m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
To validate CTP, relative to the reference standard of initial clinical assessment, for predicting poor neurological outcome (≥4 on modified Rankin scale) at hospital discharge in CCAP. | 48 hours
  The primary outcome is to check the accuracy of CTP compared to the clinical assessment in predicting the poor neurological outcome in comatose cardiac arrest patients at hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Jai Shankar, MD FRCPC, Principal Investigator — University of Manitoba
Locations (1):
- St. Boniface Hospital, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alcock S, Singh S, Wiens EJ, Singh N, Ande SR, Lampron K, Huang B, Kirkpatrick I, Trivedi A, Schaffer SA, Shankar JS. CT perfusion for Assessment of poor Neurological outcome in Comatose Cardiac Arrest Patients (CANCCAP): protocol for a prospective study. BMJ Open. 2023 Jun 2;13(6):e071166. doi: 10.1136/bmjopen-2022-071166. PMID 37270194